CLINICAL TRIAL: NCT00973713
Title: Phase II Study of RAD001 in Advanced Cholangiocarcinoma
Brief Title: Study of RAD001 in Advanced Cholangiocarcinoma: RADiChol
Acronym: RADiChol
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Austin Health (Other Government)
Responsible Party: Niall Tebbutt, Austin Health
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H2009/3522
Record Dates: First submitted 2009-09-08; First posted 2009-09-09 (Estimated); Last update posted 2009-09-09 (Estimated); Status verified 2009-09

CONDITIONS: Cholangiocarcinoma
Keywords: Advanced cholangiocarcinoma
MeSH Terms: conditions — Cholangiocarcinoma | interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- RAD001 10mg/d (Experimental)
  Interventions: Drug: RAD001

INTERVENTIONS:
Drug: RAD001 — 10mg/d
  Other Names: Everolimus

SUMMARY:
This is a clinical trial investigating the effectiveness and safety of the study drug RAD001 in patients with advanced (metastatic) cholangiocarcinoma. Palliative chemotherapy provides some benefit to this group of patients. However, chemotherapy treatment only shows low rates of radiological response and short times to tumour progression. Therefore, further treatment options are urgently required.

In laboratory studies, RAD001 has been shown to interrupt the signals that cancer cells use to grow, spread and form new blood vessels (angiogenesis). RAD001 has been approved for the treatment of kidney cancer. It has also been approved for use in Australia for the treatment of patients with kidney and liver transplants, and has been used in thousands of patients worldwide for this indication. Preliminary studies suggest that RAD001 may have activity in a range of other cancers. This study will evaluate the activity of RAD001 in advanced cholangiocarcinoma.

DETAILED DESCRIPTION:
27 patients from approximately four hospitals in Australia will participate in this trial, with approximately 15 patients being enrolled at Austin Health. All participants will receive the same treatment (RAD001 10mg/d given orally).

After screening for eligibility, participants will receive RAD001 10mg/d until tumour progression.

Participants will undergo regular CT scans (every 6 weeks during treatment) to evaluate the effectiveness of treatment. Providing they are tolerating treatment satisfactorily, they may receive study treatment until progression of disease.

Blood samples will be taken during the screening phase and every 3 weeks during the treatment phase of the trial. Participants will be followed-up every 3 months to find out about survival status, new chemotherapy or biological treatment and the outcome of any ongoing adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically/cytologically confirmed adenocarcinoma of gall bladder, intra or extra-hepatic biliary tract
2. Metastatic or locally advanced (unresectable) disease
3. Adequate organ function; creatinine<1.5xULN, BR<1.5xULN Neut>1.5, Pts>100
4. WHO Performance status 0-2
5. No prior chemotherapy for advanced Cholangiocarcinoma (Prior adjuvant chemotherapy is accepted)
6. Measurable or non-measurable disease
7. Informed consent for study participation and donation of tumour tissue for evaluation of relevant translational endpoints

Exclusion Criteria:

1. Cytotoxic chemotherapy or immunotherapy within 4 weeks prior to enrolment
2. Prior therapy with mTOR inhibitors (sirolimus, temsirolimus, everolimus)
3. Known intolerance or hypersensitivity to RAD001 (everolimus) or other rapamycins (sirolimus, temsirolimus)
4. Uncontrolled diabetes mellitus or hyperlipidaemia
5. Patients who have any severe and/or uncontrolled medical conditions
6. Active or uncontrolled severe infection
7. Cirrhosis, chronic active hepatitis or chronic persistent hepatitis
8. Severely impaired lung function
9. Patients with a known history of HIV seropositivity
10. Patients who have a history of another primary malignancy (Exceptions include non-melanoma skin cancer, carcinoma in situ of uterine cervix, or any other cancer treated with curative intent without evidence of relapse for more than 2 years)
11. Female patients who are pregnant or nursing (lactating), or adults of reproductive potential who are not using effective birth control methods. If barrier contraceptives are being used, these must be continued throughout the trial by both sexes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2009-09; Primary Completion 2011-09 (Estimated); Study Completion 2012-03 (Estimated)

PRIMARY OUTCOMES:
Tumour control | 12 weeks

SECONDARY OUTCOMES:
Overall survival | 2 years
Toxicity | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Austin Health, Melbourne, Victoria, Australia